CLINICAL TRIAL: NCT05157477
Title: Targeting the Sensory Disturbance in Autism Spectrum Disorder: The Effectiveness of Cognitive-behavior Therapy-based Virtual Reality Exposure Program
Brief Title: Targeting the Sensory Disturbance in Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201712172RINC
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Autistic Disorders Spectrum
Keywords: autism spectrum; sensory disturbance; intervention; virtual reality; cognitive behavior therapy
MeSH Terms: conditions — Child Development Disorders, Pervasive; Sensation Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-Group (Experimental): The participants who are randomized into 'CBT-based VR exposure program' (CBT+VR group) will receive the individual intervention weekly with a total of 8 sessions. The therapists, PI (Chien YL) and a clinical psychologist who is familiar with ASD psychopathology and CBT approach, will provide the CBT-based VR exposure intervention for each individual every week based on the above protocol. The participants complete the homework (i.e., relaxation and real-life exposure) between the sessions, and record 'anxiety level' before, during, and after the real-life exposure. The outcome measures will be scheduled at the end of intervention (8th week) within one week of program closure.
  Interventions: Behavioral: CBT-based VR exporsure program
- CBT-GROUP (Experimental): The 'CBT alone' intervention applies the same protocol excluding VR exposure, which is replaced by traditional role play with the therapist.
  Interventions: Behavioral: CBT-based VR exporsure program
- Control group (No Intervention): The participants who are randomized into control group will be regularly followed in a naturalistic outpatient clinic setting (every 2-4 week). During the clinic, sensory and socioemotional problems will be discussed face-to-face for 10 to 20 minutes, some self-help books will be recommended.

INTERVENTIONS:
Behavioral: CBT-based VR exporsure program — This project seeks to establish a 8-week CBT-based VR exposure program to tackle sensory problems in ASD according to the theory of exposure and desensitization (both social and non-social scenarios) as well as identifying dysfunctional thought and searching for alternative thinking. In brief, this program aims to build up the core competence of the ASD individuals in facing the sensory environment, including (1) Relaxation skills (2) Ranking the fearful sensory situations (3) Anxiety coping strategy (3) Graded exposure (4) Cognitive appraisal and restructuring: identifying the dysfunctional thought when facing the social situations and figuring out alternative thinking.
  Arms: CBT-GROUP; VR-Group

SUMMARY:
This study aims to establish a cognitive-behavior therapy (CBT) based virtual exposure (VR) exposure program to train ASD adults coping with everyday sensory scenarios. Through the practice and training, the ASD participants may learn the strategy to deal with the common sensory scenarios and master the anxiety around the exposure. The anticipatory anxiety and the maladaptive behaviors may be decreased along with the process of desensitization, while the functional impairment related to sensory sensitivity can partly be recovered.

ELIGIBILITY:
Inclusion Criteria:

* young adult aged between 18 and 45 years who had a diagnosis of ASD from a licensed mental health or medical professional based on DSM-5;
* has sensory and social problems as reported by the participant and the caregiver;
* is motivated to participate in the treatment;
* is fluent in Chinese;
* has a full-scale IQ > 70 on WAIS-IV;
* scored ≧ 26 on the caregiver-reported Autism Spectrum Quotient (AQ), indicating clinical impairment associated with ASD.

Exclusion Criteria:

* A history of major mental illness (e.g., bipolar affective disorder, schizophrenia, or psychosis) or neurological diseases;
* visual impairment and/or hearing impairment that would preclude participation in the CBT-based VR exposure program

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of heart rate | Two months, first time in the first week and second time in the last week.
  The change of heart rate is related to the activation level of sympathetic nervous system, which can describe the change on anxiety level.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No